CLINICAL TRIAL: NCT01137448
Title: The Effect of Weight Loss on Psoriasis Area Severity Index in Adult Psoriasis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The site did not have enough funds to complete study arrengments and start to enrolling. The site was not able to enroll subjects.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Adelaide Hebert, Professor, Director - Pediatric Dermatology, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5T35DK007676-18 (NIH)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Psoriasis; Obesity
Keywords: Psoriasis; Obesity
MeSH Terms: conditions — Psoriasis; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Loss (Experimental): Subjects will be enrolled in a weight loss program and will receive weight loss and nutritional counseling.
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss — Subjects will enroll in a weight loss program and participate in weight loss counseling 6 times over the course of 6 months.

SUMMARY:
The purpose of this study is to evaluate the effect that weight loss has on the severity of psoriasis in obese subjects. Fifty obese (BMI equal to or greater than 30) patients with moderate to severe plaque psoriasis will be enrolled in a weight loss intervention program. The severity of their psoriasis will be reevaluated at month 3 and month 6 of the program to determine what effect weight loss has had on their psoriasis. Serum TNF-alpha will be measured at month 0 and month 6. The hypothesis that will be tested is that weight loss will lead to a significant improvement in the severity of psoriasis and a reduction in TNF-alpha levels.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* A Body Mass Index (BMI) >/= 30
* Subject has plaque psoriasis
* A Psoriasis Area Severity Index (PASI) score >/= 10 or a total body surface area (BSA) affected by psoriasis >/= 10%
* Capable of reading, understanding, and signing a consent form
* Females of childbearing potential must have negative urine pregnancy test on Day 0, and agree to a medically effective method of birth control (as determined by the investigator)

Exclusion Criteria:

* Already participating in a study for weight loss or a study of other psoriasis treatments
* If they are on systemic therapy for their psoriasis
* Female subjects who are pregnant or planning to become pregnant
* Patients with a history of anorexia nervosa, bulimia, or other diseases that would make a weight loss program a risk to their health
* Subjects unable to comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Severity of psoriasis | 6 months
  The Psoriasis Area Severity Index (PASI) is the most common validated psoriasis severity assessment tool used in clinical trials, and combines redness, thickness, and scaliness of skin lesions with the body surface area that is affected. Most clinical trials define moderate to severe psoriasis as a PASI score of greater than or equal to 10, or a total Body Surface Area (BSA) of greater than or equal to 10%.

SECONDARY OUTCOMES:
Serum TNF-alpha levels | 6 months
  Changes in TNF-alpha levels will be correlated to weight loss. TNF-alpha levels assess inflammatory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide Hebert, MD, Principal Investigator — University of Texas Medical School - Houston
Locations (1):
- University of Texas Dermatology Clinical Research, Houston, Texas, United States